CLINICAL TRIAL: NCT00642213
Title: A Comparison of Hemorrhagic and Ischemic Strokes Among Blacks and Whites: A Population-Based Study in Cincinnati, Ohio
Brief Title: A Comparison of Hemorrhagic and Ischemic Strokes Among Blacks and Whites
Acronym: GCNKSS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Brett Kissela, Principal Investigator, University of Cincinnati
Other Study IDs: UC IRB 2013-3959; R01NS030678 (NIH)
Record Dates: First submitted 2008-03-19; First posted 2008-03-24 (Estimated); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Ischemic Stroke; TIA; Hemorrhage
Keywords: stroke; ischemic; TIA; hemorrhage; incidence; case-fatality; risk factors; genetic
MeSH Terms: conditions — Ischemic Stroke; Hemorrhage; Stroke; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We have collected blood and/or buccal samples from an interviewed cohort during years 1999,2005, and 2010.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ischemic stroke sample with DNA: We prospectively collected 450(1999), 502(2005), and 512(2010) ischemic stroke patients who agreed to participate and also most provided a sample for DNA. The cohort data consists of a baseline interview, medical record abstraction and various timeframes of followup interviews from 3 months to 3 years. See website (www.gcnkss.com for data forms)
- stroke data from medical record review: The second part of the study is a retrospective medical record review of all potential ischemic strokes, TIAs, and Hemorrhagic strokes in our 5 county region that occurred in all study years.

SUMMARY:
Our primary goal is to study temporal trends in the incidence rate, causes, treatment, and outcome of stroke among a large biracial metropolitan population of 1,349,351, of whom 215,611 (15%) are black (2000 Census). Such data are critical for the planning, intervention, and evaluation of public health efforts to decrease the mortality and morbidity due to stroke in the United States.

We have completed this goal for 1993-94, 1999, 2005, 2010 and 2015. We are in the process of collecting this data for 2020. In the 2020 study period we will also be ascertaining 3 year recurrence rates for all incident stroke events.

DETAILED DESCRIPTION:
For calendar years 1993-94, 1999, 2005, 2010, 2015, and 2020 we will or have identified every hospitalized or autopsied stroke and transient ischemic attack (TIA) at all regional hospitals in our region. We will also estimate the number of non-hospitalized strokes and TIAs by screening for potential cases at more than 100 outpatient sites throughout five counties in Greater Cincinnati/Northern Kentucky. We plan to identify and abstract detailed information from the medical record for every potential case. These results will be compared with data from all stroke patients identified by similar methodology in all study periods.

In addition, we have interviewed 1500 ischemic stroke patients and/or their families in the study periods 1999-2010 to obtain detailed information including demographic information, functional outcome and quality of life, access to and type of rehabilitation therapy, social support, caregiver availability and health status, access to post-hospital care, health insurance status, current health status, medications, prior risk factors, and knowledge about stroke signs and symptoms. We also obtained genetic material via a blood sample for most of this cohort.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke
* occurred in 1999/2005/2010
* >18 years old
* resides in 5 county region

Exclusion Criteria:

* <18 years old
* resides outside 5 county region
* inability to consent or have legal proxy consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort:Ischemic stroke patient in 1999/2005/2010 that resides in the GCNK area.
  Retrospective cohorts: All stroke and TIA events occurring during the following study periods: 1993-94, 1999, 2005, 2010, 2015 and 2020. This group is ALL stroke patients of any age that resides in our 5 county region.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 1993-07; Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
mRS | discharge or 30 days
  modified Rankin Scale

SECONDARY OUTCOMES:
mortality | 1 year
  entire patient population checked for possible death record via NDI/CDC

OTHER OUTCOMES:
2020 Stroke population mRS | 3 month, 6 month, and 1 year
  we will collect 3 months, 6 months, and 1 year mRS outcomes on the 2020 stroke patients

CONTACTS AND LOCATIONS:
Overall Officials: Brett M Kissela, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
we have a website: https://www.gcnkss.com where de-identified data can be requested via an approval process
Supporting Information: Study Protocol
Time Frame: Current study data through 2015 is available via website. 2020 data will be available at a future date.
Access Criteria: please see website below
URL: https://www.gcnkss.com

REFERENCES:
- [Derived] Gillard PJ, Sucharew H, Kleindorfer D, Belagaje S, Varon S, Alwell K, Moomaw CJ, Woo D, Khatri P, Flaherty ML, Adeoye O, Ferioli S, Kissela B. The negative impact of spasticity on the health-related quality of life of stroke survivors: a longitudinal cohort study. Health Qual Life Outcomes. 2015 Sep 29;13:159. doi: 10.1186/s12955-015-0340-3. PMID 26415945